CLINICAL TRIAL: NCT02847598
Title: A 2-Part Phase 2 Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of BIIB059 in Subjects With Systemic Lupus Erythematosus and Active Skin Manifestations and in Subjects With Active Cutaneous Lupus Erythematosus With or Without Systemic Manifestations
Brief Title: Study to Evaluate BIIB059 (Litifilimab) in Cutaneous Lupus Erythematosus (CLE) With or Without Systemic Lupus Erythematosus (SLE)
Acronym: LILAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 230LE201; 2015-004359-32 (EudraCT Number)
Record Dates: First submitted 2016-06-06; First posted 2016-07-28 (Estimated); Results first posted 2023-05-15 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Systemic Lupus Erythematosus; Active Cutaneous Lupus Erythematosus
Keywords: CLE, SLE, Cutaneous Lupus Erythematosus, Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part A: BIIB059 450 mg (Experimental): BIIB059 450 mg administered SC, Q4W with an additional dose at Week 2 for a total of 7 doses (Weeks 0, 2, 4, 8, 12, 16, and 20) in participants with SLE with active skin manifestations and joint involvement.
  Interventions: Drug: BIIB059 (litifilimab)
- Part A: Placebo (Placebo Comparator): BIIB059 matching placebo administered SC, Q4W with an additional dose at Week 2 for total of 7 doses (Weeks 0, 2, 4, 8, 12, 16, and 20) in participants with SLE with active skin manifestations and joint involvement.
  Interventions: Drug: Placebo
- Part B: BIIB059 50 mg (Experimental): BIIB059 50 mg administered SC, Q4W with an additional loading dose at Week 2 for a total of 5 doses (Weeks 0, 2, 4, 8, and 12) in participants with active CLE with or without systemic manifestations.
  Interventions: Drug: BIIB059 (litifilimab)
- Part B: BIIB059 150 mg (Experimental): BIIB059 150 mg administered SC, Q4W with an additional loading dose at Week 2 for a total of 5 doses (Weeks 0, 2, 4, 8, and 12) in participants with active CLE with or without systemic manifestations.
  Interventions: Drug: BIIB059 (litifilimab)
- Part B: BIIB059 450 mg (Experimental): BIIB059 450 mg administered, Q4W with an additional loading dose at Week 2 for a total of 5 doses (Weeks 0, 2, 4, 8, and 12) in participants with active CLE with or without systemic manifestations.
  Interventions: Drug: BIIB059 (litifilimab)
- Part B: Placebo (Placebo Comparator): BIIB059 matching placebo administered SC, Q4W with an additional loading dose at Week 2 for a total of 5 doses (Weeks 0, 2, 4, 8, and 12) in participants with active CLE with or without systemic manifestations.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB059 (litifilimab) — Administered as specified in the treatment arm.
  Other Names: litifilimab
  Arms: Part A: BIIB059 450 mg; Part B: BIIB059 150 mg; Part B: BIIB059 450 mg; Part B: BIIB059 50 mg
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the efficacy of BIIB059 (litifilimab) in reducing disease activity in participants with systemic lupus erythematosus (SLE) with active cutaneous manifestations and joint involvement (Part A), and in participants with active cutaneous lupus erythematosus (CLE) (Subacute cutaneous lupus erythematosus (SCLE) or chronic CLE, including discoid lupus erythematosus (DLE)) with or without systemic manifestations (Part B). The secondary objective is to evaluate additional efficacy parameters of BIIB059 in reducing SLE/CLE disease activity, pharmacokinetic parameters, safety and tolerability of BIIB059 (Parts A and B).

ELIGIBILITY:
Key Inclusion Criteria:

Part A:

1. Diagnosis of systemic lupus erythematosus (SLE) fulfilling at least 4 out of 11 of the 1997 revised American College of Rheumatology (ACR) classification criteria for SLE along with active skin manifestations and joint involvement.
2. At least 4 tender joints and at least 4 swollen joints with at least 4 of the swollen joints in the proximal interphalangeal (PIP) joints, metacarpophalangeal (MCP) joints and/or wrist.
3. Demonstrate at least one sign of active lupus skin disease, including acute cutaneous lupus erythematosus (ACLE), subacute cutaneous lupus erythematosus (SCLE), and/or chronic cutaneous lupus erythematosus (CCLE) (e.g., discoid lupus erythematosus (DLE)), with skin activity defined by SLE Disease Activity Index 2000 (SLEDAI-2K) at the time of Screening and randomization.

Part B:

1. Active skin manifestations Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) ≥8)) and a diagnosis of cutaneous lupus erythematosus (CLE) that has been histologically confirmed (in the past or at Screening), with or without SLE manifestations.

Key Exclusion Criteria:

1. Active lupus nephritis or moderate-to-severe or chronic kidney disease.
2. Any active skin conditions other than CLE that may interfere with the study (e.g., psoriasis, non-LE skin lupus, drug-induced lupus).
3. History of chronic, recurrent (3 or more of the same type of infection in a 12-month period), or recent serious infection (e.g., pneumonia, septicemia, herpes zoster) as determined by the Investigator and requiring anti-infective treatment within 12 weeks prior to Screening.
4. Use of immunosuppressive or disease-modifying treatments for SLE or CLE that were initiated less than 12 weeks prior to Randomization.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2016-10-20 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (109):
- United States (53):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Arizona Arthritis & Rheumatology, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - TriWest Research Associates, LLC, El Cajon, California
  - Tien Q Nguyen MD Inc, Fountain Valley, California
  - MD Med Corp, Hemet, California
  - Universtiy of California, Irvine, Irvine, California
  - The Regents of the University of California, La Jolla, California
  - Purushotham Akther & Rosan Kotha, MD Inc., La Mesa, California
  - Dermatology Reserach Associates, Los Angeles, California
  - University Clinical Trials, San Diego, California
  - Richard Barthel, MD, Santa Barbara, California
  - Robin K. Dore, MD, Inc., Tustin, California
  - Inland Rheumatology Clinical Trials Inc., Upland, California
  - Nazanin Firooz, MD Inc., West Hills, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Clinical Research of West Florida- Corporate, Clearwater, Florida
  - Medical Research Center Of Miami, Miami, Florida
  - Lakes Research, LLC, Miami Lakes, Florida
  - Omega Research Consultants, Orlando, Florida
  - Compass Research, LLC, Orlando, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Advanced Medical Reserarch, PC, Sandy Springs, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Davis Group, LTD, Las Vegas, Nevada
  - Valley Hospital, Ridgewood, New Jersey
  - Institute for Rheumatic & Autoimmune diseases, Overlook Medical Center, Summit, New Jersey
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - North Shore/Long Island Jewish PRIME, Great Neck, New York
  - Univeristy of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - American Health Research, Inc., Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Ohio State University Clinical Trials, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - UPMC Arthritis Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Low Country Rheumatology, PA, North Charleston, South Carolina
  - University of Tennessee Health Sciences Center, Memphis, Tennessee
  - Austin Regional Clinic, P.A., Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Accurate Clinical Research, Inc., Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Virginia Clinical Research, Norfolk, Virginia
- Argentina (7):
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Bueno Aires, Ciudad Autonoma Bueno Aires
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, San Juan
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Shumen
  - Research Site, Sofia
- Colombia (4):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bucaramanga
  - Research Site, Medellín
- Israel (2):
  - Research Site, Jerusalem
  - Research Site, Ramat Gan
- Mexico (9):
  - Research Site, Saltillo, Coahuila
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Morelia, Michoacán
  - Research Site, Cuernavaca, Morelos
  - Research Site, Monterrey, Neuvo Leon
  - Research Site, San Luis Potosí City, San Luis Potos
  - Research Site, Mérida, Yucatán
  - Research Site, Durango
- Philippines (9):
  - Research Site, Angeles City, Pampanga
  - Research Site, Batangas
  - Research Site, Cebu City
  - Research Site, Dasmariñas
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Makati City
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Wroclaw
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Niška Banja
  - Research Site, Šabac
- South Korea (2):
  - Research Site, Suwon, Gyeonggi-do
  - Research Site, Daejeon
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Hat Yai, Changwat Songkhla
  - Research Site, Pathum Thani, Klongluang
  - Research Site, Chiang Mai, Muang
  - Research Site, Khon Kaen, Muang
  - Research Site, Bangkok, Pathumwan

REFERENCES:
- [Derived] Cho SK, Vazquez T, Werth VP. Litifilimab (BIIB059), a promising investigational drug for cutaneous lupus erythematosus. Expert Opin Investig Drugs. 2023 May;32(5):345-353. doi: 10.1080/13543784.2023.2212154. Epub 2023 May 15. PMID 37148249
- [Derived] Furie RA, van Vollenhoven RF, Kalunian K, Navarra S, Romero-Diaz J, Werth VP, Huang X, Clark G, Carroll H, Meyers A, Musselli C, Barbey C, Franchimont N; LILAC Trial Investigators. Trial of Anti-BDCA2 Antibody Litifilimab for Systemic Lupus Erythematosus. N Engl J Med. 2022 Sep 8;387(10):894-904. doi: 10.1056/NEJMoa2118025. PMID 36069871
- [Derived] Werth VP, Furie RA, Romero-Diaz J, Navarra S, Kalunian K, van Vollenhoven RF, Nyberg F, Kaffenberger BH, Sheikh SZ, Radunovic G, Huang X, Clark G, Carroll H, Naik H, Gaudreault F, Meyers A, Barbey C, Musselli C, Franchimont N; LILAC Trial Investigators. Trial of Anti-BDCA2 Antibody Litifilimab for Cutaneous Lupus Erythematosus. N Engl J Med. 2022 Jul 28;387(4):321-331. doi: 10.1056/NEJMoa2118024. PMID 35939578
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- [Derived] Hartmann S, Biliouris K, Naik H, Rabah D, Stevenson L, Shen C, Nestorov IA, Lesko LJ, Trame MN. A clinical population pharmacokinetic/pharmacodynamic model for BIIB059, a monoclonal antibody for the treatment of systemic and cutaneous lupus erythematosus. J Pharmacokinet Pharmacodyn. 2020 Jun;47(3):255-266. doi: 10.1007/s10928-020-09688-y. Epub 2020 Apr 25. PMID 32335844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 129 investigative sites in Argentina, Bulgaria, Colombia, Israel, Korea, Mexico, Philippines, Poland, Serbia, Taiwan, Thailand, and the United States from October 20, 2016 to November 18, 2019.
Pre-assignment Details: A total of 264 participants were enrolled in the study. The study had two parts, Part A (participants with Systemic lupus erythematosus (SLE) with active skin manifestations and joint involvement) and Part B (participants with active cutaneous lupus erythematosus (CLE), including discoid lupus erythematosus (DLE), with or without SLE).
Groups:
- Part A: Placebo: Participants with systemic lupus erythematosus (SLE) with active skin manifestations and joint involvement received BIIB059 matching placebo subcutaneously (SC) every 4 weeks, starting Week 0 with an additional dose at Week 2 for a total of 7 doses up to Week 20.
- Part A: BIIB059 50 mg: Participants with SLE with active skin manifestations received BIIB059 50 mg (milligrams), SC every 4 weeks, starting Week 0 with an additional dose at Week 2 for a total of 7 doses up to Week 20.
- Part A: BIIB059 150 mg: Participants with SLE with active skin manifestations received BIIB059 150 mg, SC every 4 weeks, starting Week 0 with an additional dose at Week 2 for a total of 7 doses up to Week 20.
- Part A: BIIB059 450 mg: Participants with SLE with active skin manifestations and joint involvement received BIIB059 450 mg, SC every 4 weeks, starting Week 0 with an additional dose at Week 2 for a total of 7 doses up to Week 20.
- Part B: Placebo: Participants with active cutaneous lupus erythematosus (CLE) with or without systemic manifestations received BIIB059 matching placebo administered SC every 4 weeks, starting Week 0 with an additional loading dose at Week 2 for a total of 5 doses up to Week 12.
- Part B: BIIB059 50 mg: Participants with active CLE with or without systemic manifestations received BIIB059 50 mg, SC every 4 weeks, starting Week 0 with an additional loading dose at Week 2 for a total of 5 doses up to Week 12.
- Part B: BIIB059 150 mg: Participants with active CLE with or without systemic manifestations received BIIB059 150 mg, SC every 4 weeks, starting Week 0 with an additional loading dose at Week 2 for a total of 5 doses up to Week 12.
- Part B: BIIB059 450 mg: Participants with active CLE with or without systemic manifestations received BIIB059 450 mg, SC every 4 weeks, starting Week 0 with an additional loading dose at Week 2 for a total of 5 doses up to Week 12.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Started | 56 | 6 | 6 | 64 | 33 | 26 | 25 | 48
Completed | 51 | 6 | 6 | 60 | 30 | 23 | 23 | 44
Not Completed | 5 | 0 | 0 | 4 | 3 | 3 | 2 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Consent withdrawn | 2 | 0 | 0 | 4 | 3 | 2 | 1 | 3
Not completed — Death | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (MITT) population included all randomized participants who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg | Total
Number analyzed (Participants) | 56 | 6 | 6 | 64 | 33 | 26 | 25 | 48 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.2) | 35.0 (14.4) | 40.8 (13.4) | 40.3 (11.4) | 43.4 (11.6) | 43.3 (15.3) | 43.6 (12.1) | 44.0 (12.6) | 42.1 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 6 | 5 | 63 | 30 | 20 | 20 | 36 | 229
  Male | 7 | 0 | 1 | 1 | 3 | 6 | 5 | 12 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 1 | 2 | 24 | 3 | 5 | 1 | 4 | 65
  Not Hispanic or Latino | 16 | 4 | 3 | 20 | 22 | 14 | 13 | 34 | 126
  Unknown or Not Reported | 15 | 1 | 1 | 20 | 8 | 7 | 11 | 10 | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 13
  Asian | 13 | 4 | 2 | 12 | 14 | 7 | 6 | 17 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 6 | 2 | 5 | 2 | 5 | 20
  White | 16 | 1 | 1 | 17 | 9 | 4 | 6 | 13 | 67
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 19 | 1 | 3 | 24 | 8 | 10 | 11 | 13 | 89

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Active Joint Count (28-joint Assessment) to Week 24
Description: An active joint is defined as a joint with pain and signs of inflammation (e.g., tenderness, swelling or effusion). The 28 Joint Count includes assessment of swelling and tenderness in the shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints and knees. The investigator counts how many of the 28 joints are swollen or tender at the given week.
Time Frame: Baseline to Week 24
Population: MITT population included all randomized participants in Part A who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol). Here, "number of participants analyzed" signifies number of participants analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: joints
Groups:
- Part A: Placebo: Participants with SLE with active skin manifestations and joint involvement received BIIB059 matching placebo SC every 4 weeks, starting at Week 0 with an additional dose at Week 2 for a total of 7 doses up to Week 20.
- Part A: BIIB059 450 mg: Participants with SLE with active skin manifestations and joint involvement received BIIB059 450 mg, SC every 4 weeks, starting Week 0 with an additional loading dose at Week 2 for a total of 7 doses up to Week 20.
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 41 | 2 | 1 | 52
joints | -12.7 (10.3) | -9.0 (5.7) | -13.0 (NA) — Since only 1 participant was analyzed, standard deviation (SD) was not evaluated. | -14.5 (8.7)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: BIIB059 450 mg; A Mixed Effect Model Repeat Measurement (MMRM) model is performed, using treatment group, study visit, baseline corticosteroid usage level (<=10 mg, >10 mg), region, study visit-by-treatment interaction, baseline value of the outcome measure, and baseline-by-visit interaction as fixed effect covariates. Statistical analysis for placebo and BIIB059 450 mg was planned and reported; Test type: Superiority; p = 0.037, MMRM; Least squares (LS) mean Difference = -3.4, 95% CI 2-sided [-6.7 to -0.2]

2. Primary Outcome: Part B: Percent Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score to Week 16
Description: The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) is a clinical tool that quantifies disease activity and damage in cutaneous lupus erythematosus (CLE). The activity scale (CLASI-A) includes measurements of erythema, scale and hypertrophy, and mucous membrane disease. Each part of the body is listed separately, from the scalp to the feet, in addition to sections focusing on mucous membrane involvement and alopecia. Points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Composite scores are calculated by summing the individual component scores. CLASI-A scores of 0-9, 10-20, and 21-70 represent disease severity of mild, moderate, and severe, respectively. Higher scores indicate more disease activity.
Time Frame: Baseline to Week 16
Population: MITT population included all randomized participants in Part B who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol). Here, "number of participants analyzed" signifies number of participants analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Part B: Placebo: Participants with active CLE with or without systemic manifestations received BIIB059 matching placebo administered SC every 4 weeks, starting Week 0 with an additional loading dose at Week 2 for a total of 5 doses up to Week 12.
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 31 | 23 | 24 | 42
percent change | -15.03 (37.23) | -35.52 (33.35) | -47.11 (34.10) | -41.66 (37.33)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: BIIB059 50 mg; A MMRM model is performed, using treatment group, study visit, study visit-by-treatment interaction, DLE (Yes/No), CLASI-A score (<=10 vs. >10) as fixed effect covariates; Test type: Superiority; p = 0.015, MMRM; LS mean difference = -24.29, 95% CI 2-sided [-43.70 to -4.88]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: BIIB059 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -33.42, 95% CI 2-sided [-52.71 to -14.12]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: BIIB059 450 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.001, MMRM; LS mean difference = -27.99, 95% CI 2-sided [-44.55 to -11.42]

3. Secondary Outcome: Part A : Percentage of Participants With Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity- 50 (CLASI-50) Response at Week 24
Description: CLASI-50 Response is defined as a 50% improvement from baseline in CLASI-A score at Week 24. The CLASI is a clinical tool that quantifies disease activity and damage in CLE. The activity scale (CLASI-A) includes measurements of erythema, scale and hypertrophy, and mucous membrane disease. Each part of the body is listed separately, from the scalp to the feet, in addition to sections focusing on mucous membrane involvement and alopecia. Points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Composite scores are calculated by summing the individual component scores. CLASI-A scores of 0-9, 10-20, and 21-70 represent disease severity of mild, moderate, and severe, respectively. Higher scores indicate more disease activity.
Time Frame: Week 24
Population: MITT population included all randomized participants in Part A who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol). Here, "number of participants analyzed" signifies those with baseline CLASI-A >=8 following protocol amendment.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 38 | 6 | 6 | 39
percentage of participants | 42.11 | 50 | 16.67 | 64.10

4. Secondary Outcome: Part B: Percentage of Participants With Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity- 50 (CLASI-50) Response at Week 12 and 16
Description: CLASI-50 Response is defined as a 50% improvement from baseline in CLASI-A score at Weeks 12 and 16. The CLASI is a clinical tool that quantifies disease activity and damage in CLE. The activity scale (CLASI-A) includes measurements of erythema, scale and hypertrophy, and mucous membrane disease. Each part of the body is listed separately, from the scalp to the feet, in addition to sections focusing on mucous membrane involvement and alopecia. Points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Composite scores are calculated by summing the individual component scores. CLASI-A scores of 0-9, 10-20, and 21-70 represent disease severity of mild, moderate, and severe, respectively. Higher scores indicate more disease activity.
Time Frame: Week 12, Week 16
Population: MITT population included all randomized participants in Part B who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol). Here, "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
percentage of participants
  Week 12 | 12.12 | 38.46 | 48.00 | 37.50
  Week 16: number analyzed (Participants) | 32 | 26 | 25 | 43
  Week 16 | 21.88 | 38.46 | 44.00 | 46.51

5. Secondary Outcome: Part A: Percent Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 12, 16 and 24
Description: The CLASI is a clinical tool that quantifies disease activity and damage in CLE. The activity scale (CLASI-A) includes measurements of erythema, scale and hypertrophy, and mucous membrane disease. Each part of the body is listed separately, from the scalp to the feet, in addition to sections focusing on mucous membrane involvement and alopecia. Points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Composite scores are calculated by summing the individual component scores. CLASI-A scores of 0-9, 10-20, and 21-70 represent disease severity of mild, moderate, and severe, respectively. Higher scores indicate more disease activity.
Time Frame: Baseline, Week 12, 16 and 24
Population: MITT population included all randomized participants in Part A who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol). Here, "number of participants analyzed" signifies number of participants analyzed in this outcome measure and "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 38 | 6 | 6 | 39
percent change
  Change at Week 12: number analyzed (Participants) | 37 | 6 | 6 | 38
  Change at Week 12 | -36.63 (28.23) | -29.32 (14.66) | -8.39 (34.48) | -44.36 (39.69)
  Change at Week 16: number analyzed (Participants) | 35 | 6 | 6 | 38
  Change at Week 16 | -42.55 (32.46) | -41.76 (19.72) | -6.19 (21.31) | -50.20 (38.32)
  Change at Week 24: number analyzed (Participants) | 35 | 6 | 6 | 35
  Change at Week 24 | -45.40 (34.38) | -58.61 (35.16) | -17.92 (31.16) | -60.59 (37.36)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: BIIB059 450 mg; Week 12: A MMRM model is performed, using treatment group study visit, baseline corticosteroid usage level (<=10 mg, >10 mg), region, study visit-by-treatment interaction, baseline value of the outcome measure, and baseline-by-visit interaction as fixed effect covariates. Statistical analysis for placebo and BIIB059 450 mg was planned and reported; Test type: Superiority; p = 0.220, MMRM; LS Mean Difference = -9.93, 95% CI 2-sided [-25.94 to 6.08]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: BIIB059 450 mg; Week 16: A MMRM model is performed, using treatment group (BIIB059 450 mg vs. placebo), study visit, baseline corticosteroid usage level (<=10 mg, >10 mg), region study visit-by-treatment interaction, baseline value of the endpoint, and baseline-by-visit interaction as fixed effect covariates. Statistical analysis for placebo and BIIB059 450 mg was planned and reported; Test type: Superiority; p = 0.293, MMRM; LS Mean Difference = -8.96, 95% CI 2-sided [-25.82 to 7.90]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: BIIB059 450 mg; Week 24: A MMRM model is performed, using treatment group, study visit, baseline corticosteroid usage level (<=10 mg, >10 mg), region study visit-by-treatment interaction, baseline value of the outcome measure, and baseline-by-visit interaction as fixed effect covariates. Statistical analysis for placebo and BIIB059 450 mg was planned and reported; Test type: Superiority; p = 0.062, MMRM; LS Mean Difference = -15.74, 95% CI 2-sided [-32.28 to 0.79]

6. Secondary Outcome: Part B: Percent Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 12
Description: as for outcome 5
Time Frame: Baseline, Week 12
Population: MITT population included all randomized participants in Part B who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol). Here, "number of participants analyzed" signifies number of participant analyzed in this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 32 | 23 | 24 | 44
percent change | -10.73 (34.41) | -38.72 (32.99) | -47.82 (31.80) | -35.25 (35.77)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: BIIB059 50 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.001, MMRM; LS mean difference = -30.36, 95% CI 2-sided [-48.75 to -11.97]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: BIIB059 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.001, MMRM; LS mean difference = -37.17, 95% CI 2-sided [-55.46 to -18.87]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: BIIB059 450 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.001, MMRM; LS mean difference = -26.05, 95% CI 2-sided [-41.71 to -10.40]

7. Secondary Outcome: Part A: Percentage of Participants With a >=4-point Reduction From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 24
Description: The CLASI is a clinical tool that quantifies disease activity and damage in CLE. The activity scale (CLASI-A) includes measurements of erythema, scale and hypertrophy, and mucous membrane disease. Each part of the body is listed separately, from the scalp to the feet, in addition to sections focusing on mucous membrane involvement and alopecia. Points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Composite scores are calculated by summing the individual component scores. CLASI-A scores of 0-9, 10-20, and 21-70 represent disease severity of mild, moderate, and severe, respectively. Higher scores indicate more disease activity. The percentage of participants with a >=4-point reduction from baseline in CLASI-A score are reported here.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 38 | 6 | 6 | 39
percentage of participants | 57.89 | 83.66 | 16.67 | 71.79

8. Secondary Outcome: Part B: Percentage of Participants With a >=4-point Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 12 and 16
Description: as for outcome 7
Time Frame: Week 12, Week 16
Population: MITT population included all randomized participants in Part B who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol). Here, "number of analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
percentage of participants
  Week 12 | 33.33 | 50.00 | 76.00 | 47.92
  Week 16: number analyzed (Participants) | 32 | 26 | 25 | 43
  Week 16 | 37.50 | 46.15 | 72.00 | 55.81

9. Secondary Outcome: Part A: Percentage of Participants With a >=7-point Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 24
Description: The CLASI is a clinical tool that quantifies disease activity and damage in CLE. The activity scale (CLASI-A) includes measurements of erythema, scale and hypertrophy, and mucous membrane disease. Each part of the body is listed separately, from the scalp to the feet, in addition to sections focusing on mucous membrane involvement and alopecia. Points are given for the presence of erythema, scale, mucous membrane lesions, recent hair loss, and inflammatory alopecia. Composite scores are calculated by summing the individual component scores. CLASI-A scores of 0-9, 10-20, and 21-70 represent disease severity of mild, moderate, and severe, respectively. Higher scores indicate more disease activity. The percentage of participants with a >=7-point reduction from baseline in CLASI-A score are reported here.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 38 | 6 | 6 | 39
percentage of participants | 34.21 | 66.67 | 16.67 | 56.41

10. Secondary Outcome: Part B: Percentage of Participants With a >=7-point Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) Score at Week 12 and 16
Description: as for outcome 9
Time Frame: Week 12, Week 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
percentage of participants
  Week 12 | 18.18 | 38.46 | 40.00 | 33.33
  Week 16: number analyzed (Participants) | 32 | 26 | 25 | 43
  Week 16 | 21.88 | 30.77 | 48.00 | 41.86

11. Secondary Outcome: Part A: Percentage of Participants Achieving a Systemic Lupus Erythematosus (SLE) Responder Index >=4 (SRI-4) at Week 24
Description: An SRI-4 at Week 24 was a categorical response variable (Yes/No) incorporating the following criteria for achievement of responder status (i.e., all criteria must have been met to achieve responder status): A reduction from baseline of ≥4 points in SLEDAI-2K, No new organ system affected, as defined by no new BILAG-2004 Grade A and no more than 1 new BILAG-2004 Grade B, No worsening from baseline in participant's lupus disease activity, defined by a <1-point increase in the PGA (VAS) [on a scale of 0 to 10],No changes to protocol-specified medication rules,as follows (all criteria were required to be met): No initiation or increase of SLE standard of care therapy or other disallowed concomitant therapy; Concomitant corticosteroid dosage at Week 24 to be ≤10 mg/day;Concomitant corticosteroid dosage at Week 24 was no more than at Day 1;No increase in corticosteroid dose between Weeks 17 and 24. The percentage of participants who had responded to each of the 4 criteria was also reported.
Time Frame: Week 24
Population: MITT population included all randomized participants in Part A who had received at least 1 dose of study treatment (whether or not the participants adhered to the protocol).
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 64
percentage of participants | 28.57 | 33.33 | 16.67 | 56.25

12. Secondary Outcome: Part A: Change From Baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) Score at Week 24
Description: The SLEDAI-2K is a reliable, valid, simple, 1-page activity index that measures disease activity and records features of active lupus as present or not. It uses a weighted checklist to assign a numeric score based on the presence or absence of 24 symptoms at the time of assessment or during the previous 28 days. Each symptom present is assigned between 1 and up to 8 points based on its usual clinical importance, yielding a total score that ranges from 0 points (no symptoms) to 105 points (presence of all defined symptoms), where higher scores representing increased disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 50 | 6 | 3 | 59
score on a scale | -2.1 (3.3) | -3.0 (4.7) | -1.3 (2.4) | -4.4 (4.2)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: BIIB059 450 mg; A MMRM model is performed, using treatment group, study visit, baseline corticosteroid usage level (<=10 mg, >10 mg), region, study visit-by-treatment interaction, baseline value of the outcome measure, and baseline-by-visit interaction as fixed effect covariates. Statistical analysis for placebo and BIIB059 450 mg was planned and reported; Test type: Superiority; p = 0.007, MMRM; LS Mean Difference = -1.7, 95% CI 2-sided [-3.0 to -0.5]

13. Secondary Outcome: Part A: Percentage of Participants With no New Organ System Affected at Week 24
Description: No new organ system affected, as defined by no new British Isles Lupus Activity Group (BILAG)-2004 A and no more than one new BILAG-2004 B. The BILAG-2004 index categorizes disease activity in each organ system into five different levels from A to E. Grade A represents very active disease, Grade B represents moderate disease activity, Grade C indicates mild stable disease, and grade D implies no disease activity, but suggests the organ system had previously been affected. Grade E indicates no current or previous disease activity. A score is applied to each grade of each organ system using coding scheme of A=12, B=8, C=1, and D/E=0 and is summarized as a total score ranging 0-108. Higher scores indicate more severe disease activity.
Time Frame: Week 24
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 64
percentage of participants | 82.14 | 100.00 | 50.00 | 85.94

14. Secondary Outcome: Part A: Change From Baseline in Physician's Global Assessment (PGA) of SLE Visual Analog Scale (VAS) Score at Week 24
Description: The PGA is used to quantify disease activity and is measured using an anchored VAS. The PGA asks the Investigator to assess the participants current disease activity from a score of 0 (none) to 3 (severe), where higher score means severe SLE disease activity.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 49 | 6 | 6 | 57
score on a scale | -2.46 (2.13) | -2.05 (1.18) | -0.12 (1.48) | -2.45 (2.33)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: BIIB059 450 mg; A MMRM model is performed, using treatment group (BIIB059 450 mg vs. placebo), study visit, baseline corticosteroid usage level (<=10 mg, >10 mg), region, study visit-by-treatment interaction, baseline value of the endpoint, and baseline-by-visit interaction as fixed effect covariates. Statistical analysis for placebo and BIIB059 450 mg was planned and reported; Test type: Superiority; p = 0.667, MMRM; LS mean difference = -0.16, 95% CI 2-sided [-0.90 to 0.58]

15. Secondary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose: Results in death; in the view of the Investigator, places the participant at immediate risk of death (a life-threatening event); however, this does not include an event that, had it occurred in a more severe form, might have caused death; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect.
Time Frame: Baseline up to Week 36
Population: Safety population included all the randomized participants in Part A who had received at least one dose of randomized study treatment and was based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 64
Participants
  AEs | 38 | 3 | 6 | 36
  SAEs | 6 | 0 | 1 | 3

16. Secondary Outcome: Part B: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: as for outcome 15
Time Frame: Baseline up to Week 28
Population: Safety population included all the randomized participants in Part B who had received at least one dose of randomized study treatment and was based on the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
Participants
  AEs | 22 | 18 | 15 | 38
  SAEs | 3 | 1 | 3 | 3

17. Secondary Outcome: Part A: Number of Participants With Clinically Significant Laboratory Assessment Abnormalities
Time Frame: Baseline up to Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 64
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Part B: Number of Participants With Clinically Significant Laboratory Assessment Abnormalities
Time Frame: Baseline up to Week 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
Participants | 0 | 0 | 0 | 0

19. Secondary Outcome: Part A: Number of Participants With Clinically Significant Vital Sign Abnormalities
Time Frame: Baseline up to Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 64
Participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Part B: Number of Participants With Clinically Significant Vital Sign Abnormalities
Time Frame: Baseline up to Week 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Part A: Number of Participants With Clinically Significant 12-Lead Electrocardiograms (ECGs) Abnormalities
Time Frame: Baseline up to Week 36
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 5 | 64
Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Part B: Number of Participants With Clinically Significant 12-Lead Electrocardiograms (ECGs) Abnormalities
Time Frame: Baseline up to Week 28
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
Participants | 0 | 0 | 0 | 0

23. Secondary Outcome: Part A: Number of Participants With Positive BIIB059 Antibodies
Time Frame: Baseline up to Week 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 63
Participants | 1 | 0 | 0 | 5

24. Secondary Outcome: Part B: Number of Participants With Positive BIIB059 Antibodies
Time Frame: Baseline up to Week 16
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 32 | 26 | 25 | 48
Participants | 0 | 5 | 4 | 5

25. Secondary Outcome: Part A: Absolute Change From Baseline Over Time in Immunoglobulin Levels
Time Frame: Baseline up to Week 24
Population: Safety population included all the randomized participants in Part A who had received at least one dose of randomized study treatment and was based on the actual treatment received. Here, "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: grams per Liter (g/L)
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 64
grams per Liter (g/L)
  Immunoglobulin A (IgA): Baseline | 3.350 (1.862) | 3.610 (0.730) | 4.080 (1.537) | 3.116 (1.682)
  IgA: Change at Week 16: number analyzed (Participants) | 45 | 0 | 0 | 54
  IgA: Change at Week 16 | 0.033 (0.529) |  |  | -0.006 (0.305)
  IgA: Change at Week 24: number analyzed (Participants) | 52 | 6 | 6 | 59
  IgA: Change at Week 24 | -0.093 (0.704) | -0.433 (1.188) | -0.057 (0.966) | 0.012 (0.505)
  Immunoglobulin G (IgG): Baseline | 14.423 (4.927) | 15.723 (1.584) | 17.620 (5.502) | 14.792 (6.778)
  IgG: Change at Week 16: number analyzed (Participants) | 45 | 0 | 0 | 54
  IgG: Change at Week 16 | 1.057 (2.832) |  |  | 0.233 (2.478)
  IgG: Change at Week 24: number analyzed (Participants) | 52 | 6 | 6 | 59
  IgG: Change at Week 24 | 0.874 (3.376) | -0.468 (1.333) | -0.790 (4.967) | 0.758 (2.599)
  Immunoglobulin M (IgM): Baseline | 1.046 (0.657) | 1.065 (0.507) | 1.242 (0.718) | 1.106 (0.953)
  IgM: Change at Week 16: number analyzed (Participants) | 45 | 0 | 0 | 54
  IgM: Change at Week 16 | 0.004 (0.137) |  |  | -0.065 (0.294)
  IgM: Change at Week 24: number analyzed (Participants) | 52 | 6 | 6 | 59
  IgM: Change at Week 24 | -0.003 (0.191) | -0.050 (0.113) | -0.150 (0.160) | -0.072 (0.409)

26. Secondary Outcome: Part B: Absolute Change From Baseline Over Time in Immunoglobulin Levels
Time Frame: Baseline up to Week 16
Population: Safety population included all the randomized participants in Part B who had received at least one dose of randomized study treatment and was based on the actual treatment received. Here, "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
g/L
  IgA: Baseline | 3.341 (1.113) | 3.873 (1.663) | 2.900 (1.705) | 3.061 (1.413)
  IgA: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 14
  IgA: Change at Week 12 | -0.029 (0.249) |  |  | -0.304 (0.711)
  IgA: Change at Week 16: number analyzed (Participants) | 25 | 25 | 25 | 30
  IgA: Change at Week 16 | -0.045 (0.432) | -0.117 (0.356) | -0.016 (0.376) | -0.076 (0.254)
  IgG: Baseline | 13.480 (4.193) | 14.087 (4.285) | 13.700 (5.397) | 14.874 (5.904)
  IgG: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 14
  IgG: Change at Week 12 | 0.120 (0.662) |  |  | -1.961 (4.312)
  IgG: Change at Week 16: number analyzed (Participants) | 25 | 25 | 25 | 30
  IgG: Change at Week 16 | 0.450 (3.366) | -0.776 (1.405) | -0.084 (3.975) | -0.064 (1.375)
  IgM: Baseline | 0.978 (0.553) | 0.880 (0.563) | 1.095 (0.656) | 0.993 (0.757)
  IgM: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 14
  IgM: Change at Week 12 | -0.009 (0.061) |  |  | -0.028 (0.096)
  IgM: Change at Week 16: number analyzed (Participants) | 25 | 25 | 25 | 30
  IgM: Change at Week 16 | -0.016 (0.125) | -0.072 (0.119) | -0.045 (0.217) | -0.035 (0.150)

27. Secondary Outcome: Part A: Absolute Change From Baseline in Vaccine Titers - Streptococcus Pneumoniae (S. Pneumoniae) at Week 24
Description: Vaccine-related immunoglobulin (Ig) titers for Pneumococcus (S. pneumoniae) were analyzed, including 23 types of serotypes (sero). AB = Antibody.
Time Frame: Baseline to Week 24
Population: Safety population included all the randomized participants in Part A who had received at least one dose of randomized study treatment and was based on the actual treatment received. Here, "overall number of participants analyzed" signifies number of participants analyzed in this outcome measure and "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 54 | 6 | 6 | 63
milligrams per liter (mg/L)
  Sero 1 IgG AB: Baseline | 2.017 (4.9787) | 3.873 (3.8400) | 2.705 (5.3558) | 1.495 (3.3589)
  Sero 1 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 1 IgG AB: Change at Week 24 | 0.445 (1.9595) | 0.055 (2.9840) | -0.565 (1.4395) | 0.475 (3.5101)
  Sero 2 IgG AB: Baseline | 1.562 (2.4661) | 5.715 (6.9239) | 4.202 (4.8105) | 1.626 (2.6861)
  Sero 2 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 2 IgG AB: Change at Week 24 | 0.014 (0.8316) | -1.648 (7.1790) | -1.975 (3.2500) | -0.011 (1.2676)
  Sero 3 IgG AB: Baseline | 1.2607 (1.77918) | 2.1450 (2.39861) | 1.2733 (0.96790) | 1.6579 (3.35454)
  Sero 3 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 3 IgG AB: Change at Week 24 | -0.0886 (0.75890) | -0.2017 (2.43817) | -0.2067 (1.39370) | 0.8122 (3.62090)
  Sero 4 IgG AB: Baseline | 0.734 (1.2954) | 2.602 (4.4908) | 1.317 (1.5754) | 0.429 (0.5696)
  Sero 4 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 4 IgG AB: Change at Week 24 | -0.025 (0.5104) | -1.510 (4.9524) | -0.795 (1.6009) | 0.060 (0.6525)
  Sero 5 IgG AB: Baseline | 4.921 (4.2218) | 10.693 (17.4616) | 13.507 (17.7231) | 4.442 (3.9255)
  Sero 5 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 5 IgG AB: Change at Week 24 | 0.813 (3.9116) | -4.692 (19.3477) | -7.322 (16.4934) | 0.329 (2.3390)
  Sero 6 IgG AB: Baseline | 3.348 (6.4940) | 4.462 (4.1178) | 4.458 (6.1968) | 1.957 (2.7845)
  Sero 6 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 6 IgG AB: Change at Week 24 | -0.448 (2.4975) | -2.168 (5.1775) | -3.083 (5.3923) | 0.070 (2.4772)
  Sero 7 IgG AB: Baseline | 6.4300 (10.99806) | 8.5333 (7.97928) | 7.0033 (8.53321) | 3.0983 (6.90958)
  Sero 7 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 7 IgG AB: Change at Week 24 | -1.0336 (5.35192) | -1.3283 (7.23188) | -2.8917 (5.30027) | 0.3053 (3.13517)
  Sero 8 IgG AB: Baseline | 3.1978 (7.08938) | 3.1933 (3.01698) | 2.6183 (3.21210) | 1.5890 (4.46616)
  Sero 8 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 8 IgG AB: Change at Week 24 | 0.0925 (1.10700) | -1.3300 (3.85666) | -1.5483 (3.27227) | 0.1281 (0.84548)
  Sero 9N IgG AB: Baseline | 1.781 (2.9291) | 2.710 (3.7028) | 2.810 (4.4518) | 2.337 (4.6658)
  Sero 9N IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 9N IgG AB: Change at Week 24 | 0.217 (1.7957) | -1.327 (3.8703) | -0.907 (2.8144) | 0.499 (4.0782)
  Sero 9V IgG AB: Baseline | 1.0274 (1.44706) | 1.8300 (3.00647) | 1.5900 (1.79117) | 2.2696 (4.71508)
  Sero 9V IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 9V IgG AB: Change at Week 24 | 0.3963 (1.70256) | -0.0767 (0.64252) | -0.5750 (1.02039) | 0.6701 (4.70300)
  Sero 10A IgG AB: Baseline | 6.443 (5.8006) | 17.847 (32.7160) | 14.040 (14.0133) | 7.631 (8.2417)
  Sero 10A IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 10A IgG AB: Change at Week 24 | 0.502 (7.1412) | -8.062 (36.3708) | 0.100 (9.5476) | -0.384 (5.8464)
  Sero 11A IgG AB: Baseline | 1.768 (1.9872) | 3.203 (3.6280) | 4.095 (4.7768) | 2.308 (3.0647)
  Sero 11A IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 11A IgG AB: Change at Week 24 | 0.241 (1.1929) | -1.615 (4.5191) | -0.782 (5.3918) | -0.276 (1.6589)
  Sero 12F IgG AB: Baseline | 0.852 (2.5002) | 2.355 (3.5388) | 2.077 (2.0373) | 0.262 (0.3381)
  Sero 12F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 12F IgG AB: Change at Week 24 | 0.060 (0.8496) | -1.648 (3.7849) | -1.220 (1.7397) | -0.072 (0.1772)
  Sero 14 IgG AB: Baseline | 7.910 (11.3177) | 13.982 (16.1988) | 8.167 (9.5488) | 5.183 (6.5611)
  Sero 14 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 14 IgG AB: Change at Week 24 | -0.635 (6.6892) | -7.027 (19.5245) | -0.798 (7.1605) | 0.597 (3.6401)
  Sero 15B IgG AB: Baseline | 3.926 (5.7931) | 6.287 (7.4576) | 4.332 (4.0216) | 3.690 (5.3754)
  Sero 15B IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 15B IgG AB: Change at Week 24 | 0.603 (5.1284) | -2.262 (9.1738) | -1.607 (4.1148) | -0.341 (2.2893)
  Sero 17F IgG AB: Baseline | 4.817 (5.7702) | 11.422 (16.0156) | 11.952 (10.2915) | 4.277 (4.8458)
  Sero 17F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 17F IgG AB: Change at Week 24 | 0.427 (4.6695) | -6.123 (17.3744) | -5.898 (9.5001) | 1.330 (4.8122)
  Sero 18C IgG AB: Baseline | 3.229 (4.8212) | 3.475 (2.2460) | 2.980 (1.8997) | 2.485 (3.8363)
  Sero 18C IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 18C IgG AB: Change at Week 24 | -0.096 (2.8194) | -1.172 (2.2061) | -0.915 (1.0038) | 0.054 (2.2468)
  Sero 19A IgG AB: Baseline | 15.2372 (11.46102) | 35.2000 (58.79083) | 50.3175 (56.06189) | 14.9554 (11.40262)
  Sero 19A IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 19A IgG AB: Change at Week 24 | 2.2418 (6.97357) | -18.0750 (61.75995) | -29.3558 (44.83082) | 4.0988 (9.00464)
  Sero 19F IgG AB: Baseline | 4.203 (6.4231) | 10.857 (14.6665) | 8.353 (8.4621) | 2.609 (3.1856)
  Sero 19F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 19F IgG AB: Change at Week 24 | 0.651 (3.5642) | -6.447 (16.0973) | -3.673 (8.5727) | 1.136 (3.2837)
  Sero 20 IgG AB: Baseline | 5.4506 (6.82628) | 26.7958 (45.54328) | 21.8742 (22.32961) | 4.0902 (4.01659)
  Sero 20 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 20 IgG AB: Change at Week 24 | 0.0455 (4.96426) | -21.4475 (46.04992) | -13.0942 (16.16771) | 1.2437 (2.42526)
  Sero 22F IgG AB: Baseline | 1.563 (2.0162) | 5.743 (10.5586) | 5.525 (6.4123) | 1.138 (1.6187)
  Sero 22F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 22F IgG AB: Change at Week 24 | 0.244 (1.8324) | -4.000 (11.1710) | -3.657 (6.6997) | 0.087 (0.9350)
  Sero 23F IgG AB: Baseline | 1.401 (2.0138) | 1.897 (1.3080) | 0.685 (0.3293) | 1.797 (2.7461)
  Sero 23F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 23F IgG AB: Change at Week 24 | 0.078 (1.0468) | -0.150 (1.3425) | 0.190 (0.4725) | 0.125 (1.8192)
  Sero 33F IgG AB: Baseline | 2.610 (4.4802) | 6.600 (12.2931) | 5.630 (5.3371) | 1.800 (2.2552)
  Sero 33F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 33F IgG AB: Change at Week 24 | -0.392 (1.7998) | -5.042 (12.7997) | -3.740 (4.4122) | 0.066 (1.1380)

28. Secondary Outcome: Part B: Absolute Change From Baseline in Vaccine Titers - Streptococcus Pneumoniae (S. Pneumoniae) at Week 12
Description: as for outcome 27
Time Frame: Baseline to Week 12
Population: Safety population included all the randomized participants in Part B who had received at least one dose of randomized study treatment and was based on the actual treatment received. Here, "overall number of participants analyzed" signifies number of participants analyzed in this outcome measure and "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 10 | 1 | 0 | 21
mg/L
  Sero 1 IgG AB: Baseline | 3.538 (6.0374) | 0.210 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 1.930 (2.6639)
  Sero 1 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 1 IgG AB: Change at Week 12 | 4.193 (9.8131) |  |  | 0.116 (0.4689)
  Sero 2 IgG AB: Baseline | 4.7775 (10.24616) | 0.9900 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 3.9669 (8.68701)
  Sero 2 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 2 IgG AB: Change at Week 12 | -0.4586 (0.72158) |  |  | -0.4734 (4.04649)
  Sero 3 IgG AB: Baseline | 3.881 (7.0122) | 0.400 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 1.133 (1.0457)
  Sero 3 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 3 IgG AB: Change at Week 12 | -1.886 (5.4670) |  |  | 0.307 (0.7307)
  Sero 4 IgG AB: Baseline | 3.6185 (8.92846) | 0.1000 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 1.2376 (1.90643)
  Sero 4 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 4 IgG AB: Change at Week 12 | 0.0571 (0.20934) |  |  | 0.0450 (0.63581)
  Sero 5 IgG AB: Baseline | 7.2845 (10.00019) | 3.3500 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 5.0124 (5.83330)
  Sero 5 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 5 IgG AB: Change at Week 12 | 4.4443 (7.54015) |  |  | 3.4794 (5.30014)
  Sero 6B IgG AB: Baseline | 10.7965 (29.02953) | 0.3600 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 2.9210 (4.10508)
  Sero 6B IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 6B IgG AB: Change at Week 12 | 0.2943 (0.63629) |  |  | 0.2738 (1.49780)
  Sero 7F IgG AB: Baseline | 2.482 (3.0844) | 0.660 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 3.030 (2.6854)
  Sero 7F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 7F IgG AB: Change at Week 12 | 4.399 (10.6094) |  |  | 0.796 (1.8650)
  Sero 8 IgG AB: Baseline | 3.6820 (3.59284) | 0.2300 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 2.6629 (3.61369)
  Sero 8 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 8 IgG AB: Change at Week 12 | 1.5329 (4.51498) |  |  | 0.5931 (1.32472)
  Sero 9N IgG AB: Baseline | 4.1090 (6.77642) | 0.1300 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 2.0848 (2.59536)
  Sero 9N IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 9N IgG AB: Change at Week 12 | 3.3407 (8.56070) |  |  | 0.5875 (1.62657)
  Sero 9V IgG AB: Baseline | 1.104 (1.2697) | 0.070 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 1.520 (2.4346)
  Sero 9V IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 9V IgG AB: Change at Week 12 | -0.001 (0.3491) |  |  | -0.181 (0.9893)
  Sero 10A IgG AB: Baseline | 6.760 (10.6571) | 2.140 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 6.600 (9.0014)
  Sero 10A IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 10A IgG AB: Change at Week 12 | 1.833 (3.0611) |  |  | 4.696 (13.8354)
  Sero 11A IgG AB: Baseline | 2.1860 (2.85529) | 0.3500 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 3.5831 (4.19998)
  Sero 11A IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 11A IgG AB: Change at Week 12 | 0.6293 (3.04077) |  |  | 0.6431 (1.74757)
  Sero 12F IgG AB: Baseline | 2.1680 (4.29056) | 0.2700 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 1.2424 (1.21257)
  Sero 12F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 12F IgG AB: Change at Week 12 | 1.1429 (2.54387) |  |  | 0.3638 (0.72331)
  Sero 14 IgG AB: Baseline | 5.6435 (7.09870) | 8.9000 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 11.0210 (12.99039)
  Sero 14 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 14 IgG AB: Change at Week 12 | 1.3686 (5.66545) |  |  | -1.0319 (3.43469)
  Sero 15B IgG AB: Baseline | 4.717 (9.7429) | 1.430 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 3.410 (3.5117)
  Sero 15B IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 15B IgG AB: Change at Week 12 | 0.209 (0.2118) |  |  | 0.624 (1.4874)
  Sero 17F IgG AB: Baseline | 16.0005 (15.82427) | 17.4500 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 6.8752 (9.02378)
  Sero 17F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 17F IgG AB: Change at Week 12 | -2.0357 (4.29278) |  |  | 1.4531 (3.87924)
  Sero 18C IgG AB: Baseline | 4.083 (6.6047) | 0.140 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 5.630 (7.8627)
  Sero 18C IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 18C IgG AB: Change at Week 12 | 8.439 (21.2741) |  |  | 0.077 (1.0131)
  Sero 19A IgG AB: Baseline | 24.5485 (44.24043) | 13.7700 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 16.5624 (15.27894)
  Sero 19A IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 19A IgG AB: Change at Week 12 | 3.4457 (6.31401) |  |  | 5.3575 (8.84223)
  Sero 19F IgG AB: Baseline | 4.1040 (5.50276) | 2.0500 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 3.3800 (3.26583)
  Sero 19F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 19F IgG AB: Change at Week 12 | 2.3893 (4.24918) |  |  | 1.2275 (2.05550)
  Sero 20 IgG AB: Baseline | 11.5305 (18.12761) | 0.7900 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 8.2971 (8.28676)
  Sero 20 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 20 IgG AB: Change at Week 12 | -0.2271 (5.08362) |  |  | -1.6638 (6.48421)
  Sero 22F IgG AB: Baseline | 5.9930 (10.47744) | 0.6700 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 3.8002 (6.40547)
  Sero 22F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 22F IgG AB: Change at Week 12 | -1.8500 (4.69494) |  |  | 1.8431 (5.04651)
  Sero 23F IgG AB: Baseline | 1.6980 (2.81930) | 0.5600 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 1.9957 (2.72717)
  Sero 23F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 23F IgG AB: Change at Week 12 | 1.9964 (5.10312) |  |  | 0.2775 (0.60481)
  Sero 33F IgG AB: Baseline | 5.500 (8.3404) | 0.220 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 4.245 (4.6106)
  Sero 33F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 33F IgG AB: Change at Week 12 | -0.281 (0.4481) |  |  | 0.203 (1.4614)

29. Secondary Outcome: Part A: Absolute Change From Baseline in Vaccine Titers - Clostridium Tetani (C. Tetani) and Diphtheria at Week 24
Description: Vaccine-related immunoglobulin titers for tetanus and diphtheria were analyzed using international units per milliliter (IU/mL).
Time Frame: Baseline to Week 24
Population: Safety population included all randomized participants in Part A who had received at least one dose of randomized study treatment and was based on the actual treatment received. Here, "overall number of participants analyzed" signifies number of participants analyzed in this outcome measure and "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 54 | 6 | 6 | 62
IU/mL
  C. tetani IgG Antibody: Baseline | 2.46 (2.532) | 1.73 (1.660) | 2.52 (2.219) | 3.30 (3.674)
  C. tetani IgG Antibody: Change at Week 24: number analyzed (Participants) | 50 | 6 | 6 | 58
  C. tetani IgG Antibody: Change at Week 24 | -0.07 (1.975) | 0.07 (0.437) | 1.07 (2.890) | -0.70 (2.398)
  Diphtheria IgG Antibody: Baseline | 0.33 (0.511) | 0.10 (0.089) | 0.17 (0.163) | 0.33 (0.444)
  Diphtheria IgG Antibody: Change at Week 24: number analyzed (Participants) | 50 | 6 | 6 | 58
  Diphtheria IgG Antibody: Change at Week 24 | -0.06 (0.266) | -0.03 (0.082) | 0.07 (0.163) | -0.07 (0.340)

30. Secondary Outcome: Part B: Absolute Change From Baseline in Vaccine Titers - Clostridium Tetani (C. Tetani) and Diphtheria at Week 12
Description: Vaccine-related immunoglobulin titers for tetanus and diphtheria were analyzed.
Time Frame: Baseline to Week 12
Population: Safety population included all randomized participants in Part B who had received at least one dose of randomized study treatment and was based on the actual treatment received. Here, "overall number of participants analyzed" signifies number of participants analyzed in this outcome measure and "number analyzed" signifies number of participants analyzed at specific timepoint.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 10 | 1 | 0 | 21
IU/mL
  C. tetani IgG Antibody: Baseline | 4.41 (3.469) | 3.00 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 5.04 (2.910)
  C. tetani IgG Antibody: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  C. tetani IgG Antibody: Change at Week 12 | -0.61 (1.178) |  |  | 1.20 (6.948)
  Diphtheria IgG Antibody: Baseline | 0.46 (0.465) | 0.10 (NA) — Since only 1 participant was analyzed, SD was not evaluated. |  | 0.74 (1.027)
  Diphtheria IgG Antibody: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Diphtheria IgG Antibody: Change at Week 12 | -0.01 (0.146) |  |  | 0.06 (0.875)

31. Secondary Outcome: Part A: Percent Change From Baseline Over Time in Immunoglobulin Levels
Time Frame: Baseline up to Week 24
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 56 | 6 | 6 | 64
percent change
  IgA: Change at Week 16: number analyzed (Participants) | 45 | 0 | 0 | 54
  IgA: Change at Week 16 | 1.50 (11.91) |  |  | -0.53 (9.22)
  IgA: Change at Week 24: number analyzed (Participants) | 52 | 6 | 6 | 59
  IgA: Change at Week 24 | -1.51 (18.94) | -15.55 (41.08) | -0.10 (18.22) | -0.48 (12.94)
  IgG: Change at Week 16: number analyzed (Participants) | 45 | 0 | 0 | 54
  IgG: Change at Week 16 | 7.30 (16.58) |  |  | 2.63 (15.23)
  IgG: Change at Week 24: number analyzed (Participants) | 52 | 6 | 6 | 59
  IgG: Change at Week 24 | 6.86 (19.20) | -2.53 (8.52) | -5.88 (23.39) | 6.07 (16.44)
  IgM: Change at Week 16: number analyzed (Participants) | 45 | 0 | 0 | 54
  IgM: Change at Week 16 | 0.96 (11.71) |  |  | -0.73 (40.24)
  IgM: Change at Week 24: number analyzed (Participants) | 52 | 6 | 6 | 59
  IgM: Change at Week 24 | 1.86 (19.22) | -6.73 (12.57) | -14.99 (11.74) | 0.87 (45.16)

32. Secondary Outcome: Part B: Percent Change From Baseline Over Time in Immunoglobulin Levels
Time Frame: Baseline up to Week 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 33 | 26 | 25 | 48
percent change
  Ig A: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 14
  Ig A: Change at Week 12 | -1.45 (7.14) |  |  | -5.11 (14.44)
  Ig A: Change at Week 16: number analyzed (Participants) | 25 | 25 | 25 | 30
  Ig A: Change at Week 16 | -1.32 (12.92) | -1.48 (10.13) | 0.19 (14.22) | -2.98 (7.64)
  Ig G: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 14
  Ig G: Change at Week 12 | 0.63 (5.76) |  |  | -8.40 (18.97)
  Ig G: Change at Week 16: number analyzed (Participants) | 25 | 25 | 25 | 30
  Ig G: Change at Week 16 | 2.48 (19.59) | -3.84 (11.14) | 1.05 (18.28) | -0.39 (9.81)
  Ig M: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 14
  Ig M: Change at Week 12 | -1.25 (4.98) |  |  | -1.22 (18.25)
  Ig M: Change at Week 16: number analyzed (Participants) | 25 | 25 | 25 | 30
  Ig M: Change at Week 16 | -3.62 (10.84) | -7.60 (12.86) | -1.25 (22.27) | -0.57 (11.85)

33. Secondary Outcome: Part A: Percent Change From Baseline in Vaccine Titers at Week 24
Description: Vaccine-related immunoglobulin (Ig) titers for Pneumococcus (S. pneumoniae) including 23 types of serotypes (sero), tetanus and diphtheria were analyzed. AB = Antibody
Time Frame: Baseline to Week 24
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 54 | 6 | 6 | 63
percent change
  Sero 1 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 1 IgG AB: Change at Week 24 | 53.629 (206.5979) | 2.996 (56.3607) | -10.403 (40.9969) | 159.298 (788.0577)
  Sero 2 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 2 IgG AB: Change at Week 24 | -2.263 (52.3214) | 17.857 (64.1746) | -26.089 (35.2991) | 2.207 (57.5136)
  Sero 3 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 3 IgG AB: Change at Week 24 | -10.854 (34.9399) | 530.405 (1313.1947) | 16.282 (89.2804) | 51.000 (205.2211)
  Sero 4 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 4 IgG AB: Change at Week 24 | -8.039 (43.2246) | -15.385 (70.4542) | -26.435 (50.4316) | 26.481 (143.2057)
  Sero 5 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 5 IgG AB: Change at Week 24 | 13.293 (54.1115) | 81.053 (156.0747) | 2.937 (88.0683) | 23.064 (57.0094)
  Sero 6B IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 6B IgG AB: Change at Week 24 | -8.215 (36.4547) | -7.761 (68.3190) | -40.573 (28.7097) | 34.204 (179.4443)
  Sero 7F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 7F IgG AB: Change at Week 24 | -7.560 (54.4647) | 1.928 (90.5777) | -27.272 (30.2249) | 19.827 (120.4336)
  Sero 8 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 63
  Sero 8 IgG AB: Change at Week 24 | 13.540 (64.9487) | -14.917 (72.2397) | -19.919 (55.3947) | 13.552 (54.9741)
  Sero 9N IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 9N IgG AB: Change at Week 24 | 13.302 (108.1678) | 22.663 (111.5069) | 2.985 (42.6740) | 13.703 (137.0620)
  Sero 9V IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 9V IgG AB: Change at Week 24 | 32.983 (138.1448) | -3.399 (47.7558) | -13.591 (34.6936) | 56.445 (189.5817)
  Sero 10A IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 10A IgG AB: Change at Week 24 | 19.729 (111.4367) | 101.031 (168.5588) | 11.364 (51.7417) | 24.321 (83.4616)
  Sero 11A IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 11A IgG AB: Change at Week 24 | 51.134 (146.8640) | -16.656 (93.1140) | 14.976 (131.8861) | 18.956 (90.1198)
  Sero 12F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 12F IgG AB: Change at Week 24 | -4.445 (72.6724) | -5.463 (105.9311) | -41.416 (37.8396) | -11.447 (58.0173)
  Sero 14 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 14 IgG AB: Change at Week 24 | -3.087 (55.1562) | -31.375 (69.5715) | 2.213 (83.1715) | 20.278 (136.8606)
  Sero 15B IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 15B IgG AB: Change at Week 24 | 11.206 (116.7649) | 17.353 (66.5358) | -5.380 (47.4598) | 69.305 (570.5864)
  Sero 17F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 17F IgG AB: Change at Week 24 | 20.238 (90.3348) | 1.009 (53.3534) | -29.346 (51.5854) | 51.187 (152.3694)
  Sero 18C IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 18C IgG AB: Change at Week 24 | 14.720 (64.9702) | -14.827 (57.5927) | -30.608 (35.7004) | 43.454 (218.7604)
  Sero 19A IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 19A IgG AB: Change at Week 24 | 21.433 (55.0044) | 44.814 (73.1928) | -16.275 (73.1979) | 32.146 (64.1971)
  Sero 19F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 19F IgG AB: Change at Week 24 | 54.691 (114.1882) | 5.412 (83.2939) | -20.778 (54.8585) | 101.397 (221.3435)
  Sero 20 IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 20 IgG AB: Change at Week 24 | 35.202 (90.9529) | -37.641 (33.1824) | -53.328 (21.6352) | 75.407 (168.3388)
  Sero 22F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 57
  Sero 22F IgG AB: Change at Week 24 | 11.419 (127.0639) | 23.828 (108.3336) | -27.150 (51.7944) | 20.048 (139.8965)
  Sero 23F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 59
  Sero 23F IgG AB: Change at Week 24 | 0.215 (50.6348) | 18.204 (57.8187) | 35.862 (55.9954) | 22.329 (156.8530)
  Sero 33F IgG AB: Change at Week 24: number analyzed (Participants) | 51 | 6 | 6 | 58
  Sero 33F IgG AB: Change at Week 24 | 2.245 (65.7260) | -3.348 (64.8128) | -47.069 (32.3779) | 23.533 (102.5771)
  C.tetani IgG Antibody: Change at Week24: number analyzed (Participants) | 50 | 6 | 6 | 58
  C.tetani IgG Antibody: Change at Week24 | 19.517 (194.1378) | 39.032 (83.7958) | 29.887 (80.9696) | -11.895 (48.3260)
  Diphtheria IgG Antibody: Change at Week 24: number analyzed (Participants) | 37 | 4 | 4 | 44
  Diphtheria IgG Antibody: Change at Week 24 | 15.310 (141.4934) | -50.000 (70.7107) | 77.083 (156.8461) | -8.842 (52.9312)

34. Secondary Outcome: Part B: Percent Change From Baseline in Vaccine Titers at Week 12
Description: as for outcome 33
Time Frame: Baseline to Week 12
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 10 | 1 | 0 | 21
percent change
  Sero 1 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 1 IgG AB: Change at Week 12 | 16.835 (59.1269) |  |  | 4.257 (67.8533)
  Sero 2 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 2 IgG AB: Change at Week 12 | -20.725 (23.3306) |  |  | 15.437 (65.9854)
  Sero 3 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 3 IgG AB: Change at Week 12 | -3.370 (38.0473) |  |  | 40.604 (72.3862)
  Sero 4 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 4 IgG AB: Change at Week 12 | 6.349 (31.2778) |  |  | 32.033 (125.5527)
  Sero 5 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 5 IgG AB: Change at Week 12 | 39.578 (34.1628) |  |  | 68.850 (127.9989)
  Sero 6B IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 6B IgG AB: Change at Week 12 | 11.800 (36.9732) |  |  | 43.759 (97.2095)
  Sero 7F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 7F IgG AB: Change at Week 12 | 67.784 (90.5075) |  |  | 25.297 (48.3430)
  Sero 8 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 8 IgG AB: Change at Week 12 | 28.981 (76.3568) |  |  | 41.622 (84.8290)
  Sero 9N IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 9N IgG AB: Change at Week 12 | 18.274 (61.3305) |  |  | 19.616 (74.2945)
  Sero 9V IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 15
  Sero 9V IgG AB: Change at Week 12 | -7.707 (27.1098) |  |  | -0.573 (35.9671)
  Sero 10A IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 10A IgG AB: Change at Week 12 | 62.824 (94.6871) |  |  | 60.437 (145.3385)
  Sero 11A IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 11A IgG AB: Change at Week 12 | 12.392 (69.6069) |  |  | 29.295 (118.2639)
  Sero 12F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 12F IgG AB: Change at Week 12 | 21.768 (44.1688) |  |  | 62.768 (118.4103)
  Sero 14 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 14 IgG AB: Change at Week 12 | 77.551 (191.9769) |  |  | 18.059 (75.7757)
  Sero 15B IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 15B IgG AB: Change at Week 12 | 14.160 (16.8040) |  |  | 27.188 (56.4211)
  Sero 17F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 17F IgG AB: Change at Week 12 | -14.128 (20.3094) |  |  | 19.712 (69.9092)
  Sero 18C IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 18C IgG AB: Change at Week 12 | 36.970 (99.7771) |  |  | 8.882 (41.3781)
  Sero 19A IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 19A IgG AB: Change at Week 12 | 15.179 (28.0371) |  |  | 44.140 (113.5780)
  Sero 19F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 19F IgG AB: Change at Week 12 | 54.773 (49.4505) |  |  | 46.995 (90.7514)
  Sero 20 IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 20 IgG AB: Change at Week 12 | 1.131 (51.4091) |  |  | 0.714 (49.6361)
  Sero 22F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 22F IgG AB: Change at Week 12 | -14.748 (45.9399) |  |  | 38.974 (83.4963)
  Sero 23F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 23F IgG AB: Change at Week 12 | 52.210 (75.6486) |  |  | 16.859 (40.1773)
  Sero 33F IgG AB: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  Sero 33F IgG AB: Change at Week 12 | 0.600 (31.4400) |  |  | 26.241 (66.5051)
  C. tetani IgG Antibody: Change at Week 12: number analyzed (Participants) | 7 | 0 | 0 | 16
  C. tetani IgG Antibody: Change at Week 12 | -6.387 (18.2069) |  |  | 27.872 (128.3927)
  Diphtheria IgG Antibody: Change at Week 12: number analyzed (Participants) | 6 | 0 | 0 | 14
  Diphtheria IgG Antibody: Change at Week 12 | 0.000 (34.0588) |  |  | 28.845 (132.2208)

35. Secondary Outcome: Part A: Serum Concentration of BIIB059
Time Frame: Part A: pre-dose on Days 1, 29, 85 and 113 and post-dose on Days 1, 8, 29, 85, 169, 197 and 253
Population: The PK population included the safety participants who had at least 1 PK concentration measurement. The number analyzed is the number of participants with data available for analysis at the specified time point. The number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg
Number analyzed (Participants) | 6 | 6 | 64
nanogram per milliliter (ng/mL)
  Day 1: Pre-dose | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Day 1: Post-dose: number analyzed (Participants) | 6 | 5 | 51
  Day 1: Post-dose | 0.7 (0.6) | 2.1 (1.3) | 1.9 (2.1)
  Day 8: number analyzed (Participants) | 6 | 6 | 62
  Day 8 | 5.5 (2.0) | 17.1 (4.1) | 45.5 (16.5)
  Day 29: Pre-dose: number analyzed (Participants) | 6 | 6 | 61
  Day 29: Pre-dose | 7.0 (3.3) | 23.7 (7.2) | 53.6 (19.7)
  Day 29: Post-dose: number analyzed (Participants) | 6 | 5 | 60
  Day 29: Post-dose | 7.9 (4.2) | 25.9 (5.6) | 52.5 (20.5)
  Day 85: Pre-dose: number analyzed (Participants) | 6 | 6 | 59
  Day 85: Pre-dose | 3.9 (1.6) | 12.7 (3.7) | 34.7 (19.1)
  Day 85: Post-dose: number analyzed (Participants) | 0 | 0 | 52
  Day 85: Post-dose |  |  | 36.1 (23.2)
  Day 113: Pre-dose: number analyzed (Participants) | 6 | 6 | 59
  Day 113: Pre-dose | 3.4 (1.5) | 11.3 (5.2) | 34.6 (20.8)
  Day 169: number analyzed (Participants) | 6 | 4 | 59
  Day 169 | 3.7 (1.5) | 12.8 (4.8) | 32.0 (18.6)
  Day 197: number analyzed (Participants) | 4 | 4 | 56
  Day 197 | 0.9 (0.6) | 4.1 (2.3) | 12.6 (10.3)
  Day 253: number analyzed (Participants) | 0 | 1 | 38
  Day 253 |  | 0.4 (NA) — Since only 1 participant was evaluated, standard deviation was not estimable. | 2.8 (2.5)

36. Secondary Outcome: Part B: Serum Concentration of BIIB059
Time Frame: Part B: pre-dose on Days 1, 29, 85 and post-dose on Days 1, 29, 85, 113, 141, 169 and 197
Population: The PK population included the safety participants who had at least 1 PK concentration measurement. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
Number analyzed (Participants) | 26 | 25 | 48
ng/mL
  Day 1: Pre-dose: number analyzed (Participants) | 26 | 25 | 47
  Day 1: Pre-dose | 0.0 (0.1) | 0.1 (0.2) | 0.0 (0.1)
  Day 1: Post-dose: number analyzed (Participants) | 11 | 17 | 41
  Day 1: Post-dose | 0.4 (0.3) | 1.1 (1.1) | 2.9 (3.7)
  Day 8: number analyzed (Participants) | 26 | 24 | 27
  Day 8 | 6.8 (6.6) | 13.3 (6.1) | 47.8 (16.9)
  Day 29: Pre-dose: number analyzed (Participants) | 26 | 24 | 47
  Day 29: Pre-dose | 8.3 (7.1) | 16.9 (9.1) | 60.2 (23.3)
  Day 29: Post-dose: number analyzed (Participants) | 23 | 24 | 44
  Day 29: Post-dose | 8.7 (6.6) | 17.6 (10.2) | 61.0 (24.2)
  Day 85: Pre-dose: number analyzed (Participants) | 22 | 24 | 29
  Day 85: Pre-dose | 3.8 (3.4) | 11.0 (6.5) | 42.0 (17.1)
  Day 85: Post-dose: number analyzed (Participants) | 21 | 24 | 29
  Day 85: Post-dose | 4.1 (3.6) | 11.6 (5.8) | 42.0 (17.0)
  Day 113: number analyzed (Participants) | 22 | 25 | 30
  Day 113 | 4.6 (5.9) | 12.1 (6.5) | 43.2 (14.3)
  Day 141: number analyzed (Participants) | 14 | 22 | 44
  Day 141 | 2.5 (3.3) | 4.6 (3.7) | 19.3 (9.6)
  Day 169: number analyzed (Participants) | 4 | 12 | 39
  Day 169 | 2.4 (2.0) | 2.2 (1.1) | 7.4 (5.0)
  Day 197: number analyzed (Participants) | 2 | 8 | 35
  Day 197 | 0.8 (0.7) | 1.1 (0.4) | 3.4 (2.3)

ADVERSE EVENTS:
Time Frame: Part A: up to Week 36, Part B: up to Week 28
Description: Safety population included all the randomized participants in Part A and B who had received at least one dose of randomized study treatment and was based on the actual treatment received.
Groups:
- Part A: Placebo: Participants with SLE with active skin manifestations and joint involvement received BIIB059 matching placebo, SC every 4 weeks, starting Week 0 with an additional dose at Week 2 for a total of 7 doses up to Week 20.
Arm/Group | Part A: Placebo | Part A: BIIB059 50 mg | Part A: BIIB059 150 mg | Part A: BIIB059 450 mg | Part B: Placebo | Part B: BIIB059 50 mg | Part B: BIIB059 150 mg | Part B: BIIB059 450 mg
All-Cause Mortality (participants affected / at risk) | 3/56 | 0/6 | 0/6 | 0/64 | 0/33 | 0/26 | 0/25 | 0/48
Serious Adverse Events (participants affected / at risk) | 6/56 | 0/6 | 1/6 | 3/64 | 3/33 | 1/26 | 3/25 | 3/48
Other Adverse Events (participants affected / at risk) | 22/56 | 3/6 | 6/6 | 22/64 | 19/33 | 16/26 | 10/25 | 28/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=56) | Part A: BIIB059 50 mg (N=6) | Part A: BIIB059 150 mg (N=6) | Part A: BIIB059 450 mg (N=64) | Part B: Placebo (N=33) | Part B: BIIB059 50 mg (N=26) | Part B: BIIB059 150 mg (N=25) | Part B: BIIB059 450 mg (N=48)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal artery thrombosis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parasitic gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Systemic viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Skin angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=56) | Part A: BIIB059 50 mg (N=6) | Part A: BIIB059 150 mg (N=6) | Part A: BIIB059 450 mg (N=64) | Part B: Placebo (N=33) | Part B: BIIB059 50 mg (N=26) | Part B: BIIB059 150 mg (N=25) | Part B: BIIB059 450 mg (N=48)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 1
Asthenia (General disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 2
Injection site erythema (General disorders) | 0 | 0 | 1 | 2 | 1 | 3 | 2 | 4
Influenza (Infections and infestations) | 2 | 0 | 2 | 1 | 0 | 2 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 3 | 2 | 2 | 5 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 0 | 1 | 2 | 1 | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 4 | 0 | 1 | 4 | 0 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 2 | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 2
Headache (Nervous system disorders) | 8 | 1 | 1 | 1 | 3 | 6 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2 | 1 | 1 | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spigelian hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site warmth (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Repetitive strain injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT02847598/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT02847598/SAP_001.pdf